CLINICAL TRIAL: NCT00672230
Title: The Placental and Mammary Transfer of Lutein and Zeaxanthin Into the Fetus and the Breast-fed Infant
Brief Title: Dietary Lutein and the Retinopathy of Prematurity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: OHSUeirb00000403; USDA 2005-35200-16165
Record Dates: First submitted 2008-05-02; First posted 2008-05-06 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Lactation
Keywords: Lactation; Breast milk; Lutein; Lutein supplement
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lut Supp (Experimental)
  Interventions: Dietary Supplement: Lutein supplement

INTERVENTIONS:
Dietary Supplement: Lutein supplement — Subjects will be randomized to take a lutein supplement(12mg/day) lactation weeks 5-8 or to not take a lutein supplement

SUMMARY:
The clinical trial aspect of this study is the provision of a lutein supplement to lactating women and compare the amount of lutein in the milk and blood with lactating women who do not receive the lutein supplement.

DETAILED DESCRIPTION:
About one-fourth of preterm infants who weight less than 2 3/4 pounds at birth develop an eye problem. This problem occurs in the retina (back of the eye) and may result in blindness. This eye problem is called the retinopathy of prematurity(ROP). There are two yellow pigments in the retina called lutein and zeaxanthin. These pigments may protect the retina from being damaged by light. They may also protect the retina from being damaged by oxygen. These pigments are transferred from the mother to the baby. Most of this takes place during the last trimester of pregnancy. The situation could be worse if the baby receives formula. Most baby formulas do not contain lutein and zeaxanthin; breast milk does. Another worry is that breast milk may not have enough lutein and zeaxanthin if the mother does not eat enough vegetables and fruits. The purpose of this study is to measure the transfer of lutein and zeaxanthin from the mother to the baby, to measure the amount of lutein and zeaxanthin in breast milk, to find out if taking a lutein supplement will increase the amount of lutein in breast milk and to find out if dietary lutein and zeaxanthin are involved in the development of the retinopathy of prematurity (ROP).

ELIGIBILITY:
Inclusion Criteria:

* Planning to breast feed for at least 12 weeks
* Willing to be randomized to take the lutein supplement

Exclusion Criteria:

* Insufficient quantity of breast milk

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2005-08; Primary Completion 2008-09 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Breast milk lutein, mcg/dL | 4 weeks

SECONDARY OUTCOMES:
Plasma Lutein, mcg/dL | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: William E Connor, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States